CLINICAL TRIAL: NCT06950814
Title: Prognostic Impact of Adjuvant Therapy Following Surgical Resection in Primary Hepatic Sarcomatoid Carcinoma: A Retrospective Cohort Study
Brief Title: Prognostic Impact of Adjuvant Therapy in Primary Hepatic Sarcomatoid Carcinoma
Status: Recruiting | Type: Observational
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Jiwei Huang, Clinical Professor, West China Hospital
Other Study IDs: JHuang20231
Record Dates: First submitted 2025-04-22; First posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Sarcomatoid Carcinoma; Liver Cancer; Adjuvant Therapy
MeSH Terms: conditions — Carcinoma; Liver Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Primary hepatic sarcomatoid carcinoma patients who received adjuvant therapy
  Interventions: Procedure: postoperative adjuvant therapy
- Primary hepatic sarcomatoid carcinoma patients who did not receive adjuvant therapy

INTERVENTIONS:
Procedure: postoperative adjuvant therapy — Given the rarity and high aggressiveness of PHSC, there is a lack of reliable clinical evidence on whether postoperative adjuvant therapy can benefit patients, resulting in the absence of established standard guidelines.
  Groups: Primary hepatic sarcomatoid carcinoma patients who received adjuvant therapy

SUMMARY:
In recent years, researchers have conducted extensive studies on adjuvant therapy following surgical resection of liver cancer, exploring its potential benefits and seeking effective treatment strategies. Given the rarity and high aggressiveness of primary hepatic sarcomatoid carcinoma, there is a lack of reliable clinical evidence on whether postoperative adjuvant therapy can benefit patients, resulting in the absence of established standard guidelines. Therefore, we conducted a single-center retrospective study to assess the potential benefits of postoperative adjuvant therapy for patients of primary hepatic sarcomatoid carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. patients who underwent liver resection
2. patients' postoperative paraffin pathology and immunohistochemistry results were reviewed to identify those diagnosed with PHSC

Exclusion Criteria:

1. patients who received other anti-tumor treatments before surgery, such as radiofrequency ablation (RFA), transarterial chemoembolization (TACE), radiation therapy (RT), and systemic therapy;
2. patients diagnosed with other specific types of sarcomas;
3. patients with concurrent other malignancies during the course of PHSC;
4. patients who were lost to follow-up or lacked essential clinical data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The data was collected from patients who underwent liver resection and were diagnosed with PHSC pathologically. The data was collected from the division of Liver Surgery of West China Hospital, SCU from December 2018 to May 2023.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-04-05 (Actual); Primary Completion 2025-05-03 (Estimated); Study Completion 2025-05-05 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival | From December 2018 to May 2023
  Disease-free survival (DFS) was defined as the time from liver resection to disease recurrence or death from any cause.

SECONDARY OUTCOMES:
Overall survival | From December 2018 to May 2023
  Overall survival (OS) was defined as the interval from liver resection to death or the last follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No